CLINICAL TRIAL: NCT01105455
Title: The Effect of a Low Glycemic Index Diet on Blood Sugar Control in Pregnant Women at Risk for Gestational Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Thomas Wolever, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MSH REB 09-0263-E
Record Dates: First submitted 2010-04-09; First posted 2010-04-16 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Diabetes, Gestational
Keywords: Randomized clinical trial; Gestational diabetes; Carbohydrates; Glycemic index
MeSH Terms: conditions — Diabetes, Gestational | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High fiber (Placebo Comparator): High fiber carbohydrate foods with a high / medium glycemic index. Whole wheat bread and/or brown rice are provided to subjects if they wish. Subjects are provided with a list of other recommended carbohydrate foods.
  Interventions: Other: Nutrition education
- Low GI (Active Comparator): Carbohydrate foods with a low glycemic index. Low GI rice and whole grain bread provided to subjects if they wish. Subjects are provided with a list of recommended foods.
  Interventions: Other: Nutrition education

INTERVENTIONS:
Other: Nutrition education — Group nutrition classes supplemented by handouts and provision of key study foods.

SUMMARY:
Gestational diabetes mellitus (GDM) is a condition in which high blood sugar levels occur during pregnancy. GDM increases the risk of medical complications during pregnancy which may harm the mother and her baby. Since treating GDM to reduce blood sugar reduces the risk of harm, all pregnant women are screened for GDM using a glucose challenge test (GCT). We think that a diet containing low glycemic index foods could help keep blood sugar levels normal during pregnancy and therefore prevent GDM. Thus, the purpose of this study is to see if a diet containing low glycemic index foods will reduced blood sugar after the GCT and reduce the prevalence of GDM in women at high risk for the development of GDM.

ELIGIBILITY:
Inclusion Criteria:

* Attending Mt. Sinai Maternal Fetal Medicine Unit
* Any ONE of: body mass index >=25 kg/m^2
* OR age >=35 years
* OR high risk ethnicity (Asian, South Asian, Hispanic, African, Aboriginal)

Exclusion Criteria:

* Have pre-existing diabetes (type 1 or type 2) before becoming pregnant
* Acute or chronic illness which may affect carbohydrate metabolism
* Language/literacy barriers which cannot be overcome via available resources
* >16 weeks gestation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Serum glucose concentration 1hr after glucose challenge test | 26 weeks gestation

SECONDARY OUTCOMES:
GCT outcome | 26 weeks gestation
  ie. normal, borderline, abnormal
GDM outcome | 26 weeks gestation
  Presence or absence of gestational diabetes
Maternal weight | At EACH of the following times: 12, 16, 20, 24, 28, 32, 36 and 40 weeks gestation
Mode of delivery | At time of birth of baby
  Normal or cesarean section
Presence of birth trauma | At time of birth of baby
Weight of baby | At time of birth of baby
Presence of macrosomia | At time of birth of baby
presence of large for gestational age baby | At time of birth of baby
Presence of small for gestational age baby | At time of birth of baby
food frequency questionnaire | at 12 weeks and 26 weeks gestation
Acceptability of study foods | 26 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas MS Wolever, BM, BCh, PhD, Principal Investigator — University of Toronto
Locations (1):
- Mt Sinai Hospital, Toronto, Ontario, Canada